CLINICAL TRIAL: NCT05446038
Title: Feasibility, Acceptability, and Preliminary Efficacy of an Online Multifamily Guided Self-Help Family-Based Treatment (FBT) Group for Parents of Adolescents With Anorexia
Brief Title: Multifamily Guided Self-Help Family-Based Treatment (MF-GSH-FBT)
Acronym: MF-GSH-FBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Aileen Whyte, Clinical Assistant Professor, Psychiatry and Behavioral Sciences - Child & Adolescent Psychiatry and Child Development, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 62251
Record Dates: First submitted 2022-06-21; First posted 2022-07-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multifamily Guided Self-Help Family-Based Treatment (MF-GSH-FBT) (Experimental): Treatment consists of up to 12 once-weekly online group sessions, where groups are made up of parents from 4-5 different families of young people with Anorexia. Group sessions will last approximately 50-60 minutes. Prior to each group session, parents watch recorded videos about how parents can help their child with Anorexia. Only parents, and not the young person with Anorexia, attend the group sessions.
  Interventions: Behavioral: Multi-Family Guided Self-Help FBT

INTERVENTIONS:
Behavioral: Multi-Family Guided Self-Help FBT — Previous research has shown that Family-Based Treatment (FBT) is an effective treatment for Anorexia. We hope to learn whether an adaptation of Family-Based Treatment (FBT), called online Multi-Family Guided Self-Help FBT, is feasible and acceptable for families of young people with Anorexia. The 'Self-Help' aspect of the treatment consists of a series of educational videos for parents about how to help their child with Anorexia, which parents watch on an online platform. The 'Multifamily' and 'Guided' aspects of the treatment consists of weekly meetings by Zoom for a group of parents of young people with Anorexia, with a facilitator present to guide a group discussion around whether parents feel they understood the content of the videos and whether the content is helpful.

SUMMARY:
This is a study testing whether an online Multifamily Guided Self-Help Family Based Treatment (FBT) for Anorexia Nervosa in adolescents aged 12 to 17 is acceptable and useful to families. This online Multifamily Guided Self-Help version of FBT consists of 12 weekly 60-minute telemedicine groups made up of parents from 4-5 families of young people with AN, coupled with access to an online guided self-help platform over the course of 6 months. The feasibility of online Guided Self-Help Family-Based Treatment for Anorexia is unknown, and the investigators hope to identify an adequate treatment for those who do not have access to in-person FBT.

DETAILED DESCRIPTION:
Previous research has shown that Family-Based Treatment (FBT) is an effective treatment for Anorexia Nervosa. In the first Phase of FBT, parents are encouraged to take charge of the process of renourishing their child with Anorexia. Then, once the young person with Anorexia becomes better nourished and is managing to eat in a more sustainable way, the treatment moves to Phase 2. In Phase 2 of FBT, the focus is on helping parents to step back and support their child to regain their independence around eating. Once this happens, the treatment moves to Phase 3, where the family begins to move forward with their lives in a normal way, no longer focused on the eating disorder.

The investigators hope to learn whether an adaptation of FBT, called online Multi-Family Guided Self-Help FBT, is feasible and acceptable for families of young people with Anorexia.

The 'Self-Help' aspect of the treatment consists of a series of educational videos about how to help a child with Anorexia, which parents watch on an online platform. The 'Multifamily' and 'Guided' aspects of the treatment consists of weekly meetings by Zoom for a group of parents of young people with Anorexia, with a facilitator present to guide a group discussion around whether parents feel they understood the content of the videos and whether the content is helpful.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent participants are 12-17 years of age
2. Adolescent participants live with a family (some families may contain only one parent)
3. Family members fluently speak and read English and have access to a computer with internet
4. Adolescent participants meet DSM-5 criteria for AN
5. Adolescent participants' IBW above 75%
6. Adolescent participants are medically stable for outpatient treatment according to the recommended thresholds of the American Academy of Pediatrics and the Society of Adolescent Medicine

Exclusion Criteria:

1. Associated physical illness in any form that necessitates hospitalization of the adolescent with Anorexia
2. Psychotic illness in any form, mental retardation, autism, or any other mental illness in the adolescent or parents/ carers that would interfere with the use of psychotherapy.
3. Current dependence on drugs or alcohol in adolescent or parents.
4. Physical conditions (e.g. diabetes mellitus, pregnancy) in adolescent known to influence eating or weight
5. Participants and family members do not have an adequate understanding of spoken English and are not able to speak and read English in order to participate in family therapy and the assessments.
6. Current weight is less than 75% of expected weight given age and height.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Assessed through the end of recruitment (about one year)
  Number of participants enrolled in the study per month.
Number of Treatment Sessions Attended | Through end of treatment (up to approximately 4 months)
Treatment Retention Rate | Through end of treatment (up to approximately 4 months)
  The count of participants who did not stop treatment before finishing the 12-session parent groups
Treatment Acceptability as Measured by Helping Alliance Questionnaire | Through end of treatment (up to approximately 4 months)
  The Helping Alliance Questionnaire (HAQ) is an 11-item questionnaire that measures the quality of the therapist-patient relationship and will be completed by parents.
Treatment Acceptability as Measured by Therapy Suitability and Patient Expectancy questionnaire | Through end of treatment (up to approximately 4 months)
  The Therapy Suitability and Patient Expectancy (TSPE) measures perceptions of the suitability and expectancy of the treatment provided and will be rated by parents.

SECONDARY OUTCOMES:
Eating Disorder Cognitions | Baseline and EOT (up to approximately 4 months)
  Eating Disorder Examination (EDE): This is a standardized measure that measures the severity of the characteristic psychopathology of eating disorders. It is to be administered by assessor to the adolescent with Anorexia at baseline and EOT.
Expected Body Weight | Baseline and EOT (up to approximately 4 months)
  Expected Body Weight (EBW) percentages for the adolescent with Anorexia will be calculated using Center for Disease Control metrics in children and adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Whyte, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No